CLINICAL TRIAL: NCT04897607
Title: A Pilot Pragmatic RCT of a Hospital-based Precision Pharmacotherapy Smoking Cessation Program
Brief Title: Precision Pharmacotherapy Smoking Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: University of Delaware (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Scott Siegel, Director of Population Health Research, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDD# 604572; U54GM104941 (NIH); CCC# 41042 (Other: ChristianaCHS)
Record Dates: First submitted 2021-05-14; First posted 2021-05-21 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to the precision or standard care arms in a 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Plan Option 1 (Standard Care) (Active Comparator): Standard smoking cessation counseling will be offered + participant choice of nicotine patches or varenicline. Participants are also free to decline either medication.
  Interventions: Behavioral: Standard Care
- Treatment Plan Option 2 (Precision Pharmacotherapy) (Experimental): Standard smoking cessation counseling will be offered + a recommendation to take either the nicotine patch or varenicline based on the results of the NMR test. Regardless of the recommendation, it would still remain the participant's choice to be prescribed either nicotine patches or varenicline. Participants are also free to decline either medication.
  Interventions: Behavioral: Precision pharmacotherapy

INTERVENTIONS:
Behavioral: Standard Care — Participants will be advised to quit smoking and offered a choice of nicotine replacement patches or varenicline. Participants are free to decline medication.
  Arms: Treatment Plan Option 1 (Standard Care)
Behavioral: Precision pharmacotherapy — Participants will be advised to quit smoking and provided a medication recommendation on the basis of their nicotine metabolite ratio (NMR) test (i.e., nicotine replacement patches for slower metabolizers, varenicline for faster metabolizers). Participants are free to choose either medication or decline any medication.
  Arms: Treatment Plan Option 2 (Precision Pharmacotherapy)

SUMMARY:
The purpose of this study is to determine the benefits of a personalized treatment approach, compared to a non-personalized treatment approach, for smoking cessation. In other words, this study will help us know if recommending a specific medication to individual smokers will make it easier to quit smoking than simply offering an option of medications. The specific recommendation for a medication will be based on a test that measures how quickly a smoker breaks down, or metabolizes, nicotine.

DETAILED DESCRIPTION:
Promising new evidence suggests that applying a precision pharmacotherapy approach based on the nicotine metabolite ration (NMR), a commercially available, genetically-informed marker of nicotine metabolism rate can significantly improve cessation outcomes. Evidence from multiple independent studies, including a recent randomized clinical trial (RCT), demonstrates that matching slow metabolizers of nicotine with the nicotine patch and fast metabolizers of nicotine with varenicline can maximize treatment response and minimize side effects. While encouraging, a critical gap in knowledge is how to best translate a precision pharmacotherapy approach into a hospital-based smoking cessation intervention and improve cessation rates for underserved smokers. Preliminary data suggest that personalized treatment recommendations may increase smoking cessation medication uptake and effectiveness. Thus, the scientific premise of this application is that integrating a precision pharmacotherapy approach into a hospital-based smoking cessation program will increase medication uptake and effectiveness, with particular relevance for smokers from underserved communities.

ELIGIBILITY:
Inclusion Criteria:

* current smoker (5+ cigarettes/day)
* patient at the Helen F. Graham Cancer Center & Research Institute (ChristianaCare) lung/thoracic clinic

Exclusion Criteria:

* use of non-cigarette tobacco products or smoking cessation treatment
* psychiatric or other medical contraindications to receiving smoking cessation medication
* no telephone
* medical instability
* inability to communicate in English
* unable to consent due to mental status
* estimated life expectancy of <6 months
* not a Delaware resident
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Siegel, Ph.D., Principal Investigator — Christiana Care Health Services
Locations (1):
- Helen F. Graham Cancer Center & Research Institute, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Plan Option 1 (Standard Care) | Treatment Plan Option 2 (Precision Pharmacotherapy)
Started | 17 | 20
Completed | 11 | 13
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Plan Option 1 (Standard Care) | Treatment Plan Option 2 (Precision Pharmacotherapy) | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 14 | 23
  >=65 years | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.88 (7.01) | 59.42 (9.64) | 60.03 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 11 | 11 | 22
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 20 | 37
Count of Active Smokers [Count of Participants; unit: Participants] — Count of active smokers in each study arm, based on use of combustible cigarettes (self-reported as yes to active smoking), at the beginning of the study. Calculated to observe number of patients who successfully achieve smoking cessation (primary outcome).
  Participants | 17 | 20 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieve Smoking Cessation
Description: Participants will report smoking status at the final assessment. Participants who self-report smoking cessation completed a carbon monoxide reading for biochemical confirmation of smoking status. The percentage of participants who achieve smoking cessation in each arm will be evaluated.
Time Frame: 4-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Plan Option 1 (Standard Care) | Treatment Plan Option 2 (Precision Pharmacotherapy)
Number analyzed (Participants) | 17 | 20
Participants | 1 | 1

2. Secondary Outcome: Percentage of Participants Who Reported Using Smoking Cessation Medication (1-week)
Description: Participants will report whether smoking cessation medication was used at the first week follow-up. The percentage of participants who used medication in each arm will be evaluated.
Time Frame: 1-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Plan Option 1 (Standard Care) | Treatment Plan Option 2 (Precision Pharmacotherapy)
Number analyzed (Participants) | 17 | 20
Participants | 11 | 14

3. Secondary Outcome: Percentage of Participants Who Reported Using Smoking Cessation Medication (4-week)
Description: Participants will report whether smoking cessation medication was used during 4 week follow up. The percentage of participants who used medication in each arm will be evaluated.
Time Frame: 4-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Plan Option 1 (Standard Care) | Treatment Plan Option 2 (Precision Pharmacotherapy)
Number analyzed (Participants) | 17 | 20
Participants | 4 | 6

4. Secondary Outcome: Percentage of Participants Who Reported Use of a Smoking Medication That Matched Their NMR Profile
Description: Participants will report which smoking cessation medication, if any, was used. Medication usage will be classified as matching their NMR profile as follows: slower metabolizer = nicotine replacement therapy, faster metabolizer = varenicline. The percentage of participants who matched in each arm will be evaluated.
Time Frame: 1-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Plan Option 1 (Standard Care) | Treatment Plan Option 2 (Precision Pharmacotherapy)
Number analyzed (Participants) | 17 | 20
Participants | 5 | 11

ADVERSE EVENTS:
Time Frame: General recruitment began in February 2022 - December 2022 (approximately 10 months). Patients who were enrolled received an initial baseline intake survey followed by appointments one week (Week 1) and four weeks (Week 4) after beginning their medication. Patient data for adverse events were collected during the patient's entire enrollment (approximately 6 weeks).
Arm/Group | Treatment Plan Option 1 (Standard Care) | Treatment Plan Option 2 (Precision Pharmacotherapy)
All-Cause Mortality (participants affected / at risk) | 0/17 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/20
Other Adverse Events (participants affected / at risk) | 0/17 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Plan Option 1 (Standard Care) (N=17) | Treatment Plan Option 2 (Precision Pharmacotherapy) (N=20)
Pre-existing diabetes (Endocrine disorders) | 0 | 1 — Occurred on 8/15/22. Patient died from pre-existing, poorly controlled diabetes, that was determined to be unrelated to participation in the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Plan Option 1 (Standard Care) (N=17) | Treatment Plan Option 2 (Precision Pharmacotherapy) (N=20)
Nausea (Gastrointestinal disorders) | 0 | 1 — Event occurred on 9/20/22. Participant reported nausea from medication (varenicline), which is reported in more than 5% of people taking the medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT04897607/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT04897607/SAP_002.pdf
  • Informed Consent Form (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT04897607/ICF_003.pdf